CLINICAL TRIAL: NCT06990347
Title: A Retrospective Multicenter Cohort Study on the Efficacy and Safety of Inetetamab and Pyrotinib Combined With Chemotherapy for HER2-positive Metastatic Breast Cancer
Brief Title: A Study on the Efficacy and Safety of IPyC for HER2+ MBC
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Fan Wu, Associate Director, Fujian Medical University
Other Study IDs: K2024-534-01
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Inetetamab and Pyrotinib Combined with Chemotherapy — Inetetamab and Pyrotinib Combined with Chemotherapy

SUMMARY:
Between July 2020 and August 2024, 301 HER2-positive MBC patients from five tertiary centers received the regimen until disease progression or unacceptable toxicity. Efficacy endpoints included progression-free survival (PFS), objective response rate (ORR), and clinical benefit rate (CBR).

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent a biopsy of the metastatic site and were confirmed as having MBC
* patients who received inetetamab + pyrotinib + chemotherapy as metastasis therapy.

Exclusion Criteria:

* male patients or individuals with prior malignancy
* patients with prior or current enrollment in interventional clinical trials for MBC
* patients who received less than 2 cycles of treatment (6 weeks of inetetamab or 8 weeks of pyrotinib)
* patients who were lost to follow-up during the therapeutic process

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients from five centers, clinical oncology school of fujian medical university, fujian provincial hospital, the first affiliated hospital of xiamen university, zhangzhou zhengxing hospital and the third affiliated people's hospital of fujian university of traditional chinese medicine
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 2 years

SECONDARY OUTCOMES:
objective response rate (ORR) | 2 years
clinical benefit rate (CBR) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, China

IPD SHARING:
Plan to Share IPD: No